CLINICAL TRIAL: NCT02085837
Title: An Open Label Randomized Controlled Study to Compare the Impact of Patient Centered Nursing Services in Addition to a Nephrologist's Usual Patient Care With Usual Nephrologist's Care in Late Stage Chronic Kidney Disease Patients.
Brief Title: Healthy Transitions in Late Stage Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Steven Fishbane, Principal Investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-033
Record Dates: First submitted 2014-03-07; First posted 2014-03-13 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Educational Status; Medication Review

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Transitions Group (Experimental): * Additional nursing services will be provided to this group in addition to a usual care by Nephrologist.
  * Daily weight measurement and monitoring
  * Medication review
  * Universal dietary education
  * Focused advanced directive program
  * Countdown to fistula program
  Interventions: Other: Education; Other: Daily weight measurement and monitoring; Other: Universal Dietary education; Other: Medication review; Other: Focused advanced directive program; Other: Countdown to fistula program
- Usual Care Group (No Intervention): Usual care by nephrologist. No additional nursing support services will be provide to this group.

INTERVENTIONS:
Other: Education — Additional education will be provided by nurses to improve communication and reduce fragmentation of care.
  Arms: Healthy Transitions Group
Other: Daily weight measurement and monitoring — Monitor weight to avoid problems related to hypervolemia.
  Arms: Healthy Transitions Group
Other: Universal Dietary education — To improve diet and health
  Arms: Healthy Transitions Group
Other: Medication review — Medication will be reviewed by nurses to detect any discrepancies to reduce medication error.
  Arms: Healthy Transitions Group
Other: Focused advanced directive program — Education will be provided to increase awareness and encourage patients to have advanced directive.
  Arms: Healthy Transitions Group
Other: Countdown to fistula program — To reduce the number of patients starting dialysis with catheter in place, comprehensive stepwise intervention will be provided by nurses to ensure arterio-venous (AV) fistula placement in all appropriate patients, with coordinated follow up and failure recovery processes.
  Arms: Healthy Transitions Group

SUMMARY:
Improve health and outcome for people with late stage chronic kidney disease by providing patient centered nursing services in addition to a Nephrologist's routine patient care.

ELIGIBILITY:
Inclusion Criteria:

* Stage 4-5 Chronic Kidney Disease (CKD), defined as estimated glomerular filtration rate (eGFR) between 0-30 ml/minute
* 18 years of age or older

Exclusion Criteria:

* Cognitive impairment that is clinically apparent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Hospitalization rate | 18 months
  Reduction in hospitalization rate in intervention group as compare to control group.

SECONDARY OUTCOMES:
Improve hemodialysis access rates | 18 months
  Percentage of patients with AVF, AVG or catheters
Home dialysis | 18 months
  Increase choice of home dialysis as modality of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Steven Fishbane, MD, Principal Investigator — Northwell Health
Locations (1):
- Division of Kidney diseases and Hypertension, Great Neck, New York, United States